CLINICAL TRIAL: NCT04888403
Title: A Prospective Study on the Safety and Effectiveness of Toripalimab Combined With Neoadjuvant Radiotherapy and Chemotherapy in the Treatment of Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Exploring the Safety and Effectiveness of Toripalimab Combined With Neoadjuvant Radiotherapy and Chemotherapy in the Locally Advanced Esophageal Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, Feng Wang fengw010@163.com, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FQX-006
Record Dates: First submitted 2021-05-13; First posted 2021-05-17 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Locally Advanced Esophageal Squamous Cell Carcinoma
Keywords: locally advanced Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab combined with neoadjuvant radiotherapy and chemotherapy Single arm study (Experimental): Induction period:
  Toripalimab 240mg administered intravenously (IV) on Day 1 of each 21-day cycle for 1 cycles.
  Neoadjuvant radiotherapy after 2W: The radiotherapy dose is 41.4Gy, completed in 23 times, 5 times a week, using intensity-modulated radiotherapy (IMRT) or volume-modulated radiotherapy (VMAT); In the same period, albumin paclitaxel combined with nedaplatin chemotherapy: albumin paclitaxel 60mg/m2 + nedaplatin 25mg/m2, performed once a week, 5 times in total; Simultaneous immunotherapy: 240 mg of Toripalimab (PD-1 antibody), once every 3 weeks, 4 times in total; Received radical resection of esophageal cancer within 7 weeks after radiotherapy and chemotherapy.
  Interventions: Drug: Toripalimab+Nedaplatin+Albumin Paclitaxel

INTERVENTIONS:
Drug: Toripalimab+Nedaplatin+Albumin Paclitaxel — Toripalimab 240mg administered intravenously (IV) on Day 1 of each 21-day cycle for 1 cycles.
  Other Names:Toripalimab+Nedaplatin+Albumin Paclitaxel Neoadjuvant radiotherapy after 2W: The radiotherapy dose is 41.4Gy, completed in 23 times, 5 times a week, using intensity-modulated radiotherapy (IMRT) or volume-modulated radiotherapy (VMAT); In the same period, albumin paclitaxel combined with nedaplatin chemotherapy: albumin paclitaxel 60mg/m2 + nedaplatin 25mg/m2, performed once a week, 5 times in total; Simultaneous immunotherapy: 240 mg of Toripalimab (PD-1 antibody), once every 3 weeks, 4 times in total; Received radical resection of esophageal cancer within 7 weeks after radiotherapy and chemotherapy.
  Other Names:Toripalimab+Nedaplatin+Albumin Paclitaxel

SUMMARY:
The purpose of this study is to observe and evaluate the efficacy and safety of Toripalimab Combined With Neoadjuvant Radiotherapy and Chemotherapy in the Locally and Advanced Esophageal Squamous Cell Carcinoma

DETAILED DESCRIPTION:
In China, the incidence of esophageal cancer has declined in recent years, but the mortality rate has been ranked fourth. Morbidity and mortality were ranked sixth and fourth in all malignancies, respectively. Therefore, esophageal cancer has always been a major malignant tumor that threatens the health of our residents. Investigator designed a single-arm, open-label, phase II trial of Toripalimab Combined With Neoadjuvant Radiotherapy and Chemotherapy for locally advanced esophageal squamous cell carcinoma. The purpose of this study is to observe and evaluate the efficacy and safety of Toripalimab Combined With Neoadjuvant Radiotherapy and Chemotherapy for locally advanced esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age ≥18 years old and ≤70 years old; 2) Pathologically diagnosed thoracic esophageal squamous cell carcinoma (the midpoint of the upper and lower edges of the esophageal primary lesion is ≥25cm from the incisor); 3) There is no distant metastasis by imaging examination, and the esophageal cancer can be resected or potentially resectable after the expert consultation of thoracic surgery. The clinical stage is cT1-T2N1-N2/T3-4aN0-2M0 Ⅱ-IVA patients (AJCC 8th edition cTNM staging); 4) ECOG score 0-1 points; 5) Have not received anti-tumor treatment in the past; 6) Expected survival period> 6 months; 7) The main organ function meets the following criteria:

Blood routine examination meets the following criteria:

White blood cell (WBC) ≥3×109/L,Neutrophil count ≥ 1.5 x 109 / L,Platelet ≥ 75 x 109 / L,Hemoglobin ≥ 10.0 g / dL;

Liver function:

total bilirubin (TBIL) ≤ 2ULN,Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the upper limit of normal value;

Renal function:

creatinine clearance (cCr) ≥ 60 ml/min, creatinine (Cr) ≤ 1.5 upper limit of normal (ULN);

Heart function:

no heart disease or coronary heart disease, patients with heart function 1-2; The blood pressure of hypertensive patients should be controlled within the normal range by using antihypertensive drugs; 8)The fasting blood sugar of diabetic patients should be controlled at ≤8mmol/L through hypoglycemic drugs; 9)There are no other serious diseases that conflict with this plan (such as autoimmune diseases, immunodeficiency, organ transplantation or other diseases that require continuous hormone therapy); 10)No history of other malignant tumors; The patient himself agreed to participate in this clinical study and signed the "Informed Consent".

Exclusion Criteria:

* 1)The patient has previously received anti-tumor therapy (including chemotherapy, radiotherapy, surgery or immunotherapy, etc.) 2) The patient has or is expected to have an obvious risk of esophageal perforation, fistula and massive bleeding; 3) Exclude subjects who have previously suffered from other malignant tumors, unless they have achieved complete elimination at least 5 years before entering the study, and no additional treatment is required or expected during the study period (exceptions include but are not limited to basal or squamous cells) Skin cancer, superficial bladder cancer or carcinoma in situ of prostate, cervix or breast); 4)Subjects with known or suspected active autoimmune diseases. It is allowed to include type I diabetes, hypothyroidism that requires only hormone replacement therapy, skin diseases that do not require systemic treatment (eg, vitiligo, psoriasis, or hair loss), or in the absence of external triggers, it is not expected Subjects with relapsed conditions; 5)Clinically obvious cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction, unstable or severe angina pectoris, coronary artery bypass surgery, congestive heart failure, ventricular arrhythmia requiring medical intervention within 6 months before enrollment 、Left ventricular ejection fraction <50%, or other patients who are not expected to tolerate chemotherapy and radiotherapy; 6)Subjects suffering from conditions requiring systemic treatment with corticosteroids (>10 mg daily prednisone or equivalent dose) or other immunosuppressive drugs within 14 days prior to the administration of the study drug. In the absence of active autoimmune diseases, use inhaled or topical steroids and adrenal replacement steroids with an equivalent dose of> 10 mg daily prednisone; 7)Subjects with symptoms or interstitial lung diseases that may interfere with the detection or treatment of suspected drug-related lung toxicity; 8)Those who have previously received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or anti-CTLA-4 antibodies or any other antibodies or drugs that target T cell costimulation or checkpoint pathways as specific targets treatment； 9)All toxicities (except for kidney disease, neuropathy, hearing loss, hair loss, and fatigue) attributable to previous anti-cancer treatments must be restored to level 1 (NCI CTCAE 5th Edition) or baseline before the study drug is administered. Subjects with toxicity that can be attributed to previous anti-cancer treatments that are not expected to be relieved and lead to long-lasting sequelae (eg, peripheral neuropathy that occurs after platinum-containing treatment) are allowed to be included in the study. Peripheral neuropathy must be relieved to level 2 (NCI CTCAE 5th edition); 10)According to the opinion of the investigator, any serious or uncontrolled medical disease or active infection that may increase research participation, research drug administration related risks, or damage the subject's ability to receive the treatment of the trial protocol; 11)Known human immunodeficiency virus (HIV) test positive history or known suffering from acquired immunodeficiency syndrome (AIDS); 12)Subjects who received live vaccine/attenuated vaccine within 30 days after receiving the first treatment; 13)Patients with active viral hepatitis B or C viral hepatitis. Acute or chronic active hepatitis B or C infection, hepatitis B virus (HBV) DNA> 2000IU/ml or 104 copies/ml; hepatitis C virus (HCV) RNA> 103 copies/ml; hepatitis B surface antigen (HbsAg) and anti-HCV antibody positive at the same time; 14)History of allergies or hypersensitivity to study drug components, and history of severe hypersensitivity to any monoclonal antibody; 15)Other researchers evaluated those who did not meet the enrollment conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-07-20 (Estimated); Study Completion 2022-07-20 (Estimated)

PRIMARY OUTCOMES:
Pathologic Complete Response(pCR) | At time of surgery
  defined as the absence of any viable tumor at the time of surgical resection,as assessed by central and local pathology laboratory

SECONDARY OUTCOMES:
Major Patholgical Response(MPR) | At time of surgery
  defined as ≤ 10% residual viable tumor at the time of surgical resection,as assessed by central and local pathology laboratory
Disease-Free Survival | up to 2 years
  Time after R0 resection to disease recurrence or death
R0 resection rate | At time of surgery
  R0 is no residue under the microscope after excision
postoperative complications rate | up to 6months
  Complication refers to the occurrence of another or several diseases related to the treatment of this disease during the treatment of a certain disease

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Hennan, China